CLINICAL TRIAL: NCT05562206
Title: A 48hr Study to Test Feasibility of the Pacific Diabetes Technologies Continuous Glucose Monitor Infusion Set (CGMIS) Sensing Interstitial Glucose Continuously in the Immediate Vicinity of SQ Insulin Delivery in Adults With T1 Diabetes
Brief Title: CGMIS 48-hour Feasibility Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pacific Diabetes Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIP-01
Record Dates: First submitted 2022-09-26; First posted 2022-09-30 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Type1diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Study group (Experimental): All subjects using the study device
  Interventions: Device: CGMIS (Continuous Glucose Monitoring Infusion Set)

INTERVENTIONS:
Device: CGMIS (Continuous Glucose Monitoring Infusion Set) — An integrated combination CGM/insulin infusion system

SUMMARY:
This is a single center, single arm non-randomized study of 48-hour CGMIS wear duration incorporating two meal-challenge tests to explore the performance of a single insertion combined glucose-sensing insulin delivery cannula.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes, present for at least 6 months. If there is lack of clarity regarding the type of diabetes, the PI will make the final decision based on medical records.
* Age 18-75
* Currently using a Tandem T-Slim or Medtronic 523/723 or newer series insulin pump to treat their diabetes.
* Hgb A1C between 5.8 and 10%
* Willingness to follow all study procedures and to attend all clinic visits.
* Willingness to sign informed consent and HIPPA documents.

Exclusion Criteria:

* Need for MRI/CT/Diathermy during study participation
* Current use of Hydroxyurea
* History of chronic kidney disease
* Inability to read pump or CGM display due to reduced visual acuity
* History of unstable ischaemic heart disease or myocardial infarction within the last 3 months.
* History of chronic liver disease
* Active infection such as HIV or hepatitis
* Anemia defined by HCT at least 4 percentage points below lower limit of the reference range
* Dementia, Schizophrenia or other untreated mental illness
* Chronic substance abuse
* Chronic alcohol abuse
* Seizure disorder
* Major surgical operation within 30 days prior to screening
* History of bleeding disorder or treatment with anticoagulants.
* Allergy to acrylate-based skin adhesives
* Ongoing use of an investigational drug or device
* Female of childbearing potential who is pregnant or intending to become pregnant
* Diabetic ketoacidosis or hypoglycemia requiring hospitalization within the last 6 months
* Insulin resistance as defined by insulin requirement of more than 200 units per day
* Use of glucose-lowering medications other than insulin
* Need for uninterrupted treatment with acetaminophen
* Any other physical or mental condition judged by the PI as being exclusionary.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08-30 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Accuracy | First 48 hours
  Sensor accuracy as determined by mean absolute difference (MAD) for reference YSI venous blood glucose values ≤75 mg/dL and mean absolute relative difference (MARD) for reference YSI venous blood glucose values >75 mg/dL
Accuracy | First 48 hours
  • Sensor accuracy in the performance metrics described in the FDA iCGM Special Controls.

SECONDARY OUTCOMES:
Number of subjects who discontinue delivery of insulin through the device due to unexplained hyperglycemia | First 48 hours
  this will be the number of subjects who experience unexplained glycemic excursions requiring a cannula change
Results of tolerability questionnaire | First 48 hours
  A tolerability questionnaire will assess level of discomfort (none to severe), and duration.
Results of Draize scale | Firts 48 hours
  Draize scale will be used by study staff to evaluate the presence and severity of erythema and edema at the site of device use after removal.
Visual Analog Scale (VAS) for site discomfort | First 48 hours
  Subject will place a mark along a 100mm line to denote visually their perceived intensity of discomfort. Results will range from no discomfort to worst possible discomfort.

CONTACTS AND LOCATIONS:
Locations (1):
- Rainier Clinical Research Center, Renton, Washington, United States